CLINICAL TRIAL: NCT05883670
Title: Evaluate Efficacy and Safety of Serplulimab（HLX10）in Patients With Advanced, Recurrent and Metastatic Cervical Cancer：A Prospective, Multicenter, Non-interventive Real-world Study
Brief Title: Real-world Study of Serplulimab in 2L and Above Treatment of Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Beihua Kong, professor, Shandong University
Other Study IDs: ASTRUM-CC02
Record Dates: First submitted 2023-03-06; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: The medication plan is determined by gynecological oncology or oncology physician. Select the treatment plan containing serplulimab (single drug and/or combination), the other anti-tumor treatment schemes without intervention.
  The recommended dose of serplulimab is 300 mg IV, Day1 of each cycle. Apply the drug on the first day of each cycle until the disease progresses or intolerable toxicity occurs.The combined drugs is decided by the doctor.
  In this non-interventive study, do not change or interfere with the current medical treatment of the recruited patients.
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — Serplulimab will be administered by intravenous infusion at a dose of 300mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Other Names: HLX10

SUMMARY:
This study is a Prospective, Multicenter, non-interventive Real-world Study to evaluate the efficacy and safety of the treatment of Serplulimab in patients with Advanced,Recurrent and Metastatic Cervical Cancer. Approximately 118 eligible subjects are planned to be enrolled across all sites.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of study entry.
* Histologically or cytologically confirmed advanced, recurrent or metastatic cervical cancer.
* Received at least 1 prior systemic therapies in the recurrent or metastatic setting. Tumor progression or recurrence after treatment with therapy.
* ECOG performance status of 0 or 1.
* Patient must have at least one measurable disease as defined by RECIST 1.1.
* Ability to provide written and signed informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Life expectancy < 3 months
* Ongoing participation in another clinical study, or planned initiation of treatment in this study less than 14 days from the end of treatment in the previous clinical study.
* Known history of serious allergy to any active ingredie or any excipients list in monoclonal antibody.
* The patient has other factors that, in the judgment of the investigator, may lead to forced early termination of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Histologically or cytologically confirmed advanced, recurrent or metastatic cervical cancer，who received at least 1 prior systemic therapies in the recurrent or metastatic setting，tumor progression or recurrence after treatment with therapy.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective Response Rate is defined as the percentage of patients with Complete Response or Partial Response, as assessed by Response Evaluation Criteria in Solid Tumors v.1.1 criteria or immune Response Evaluation Criteria in Solid Tumors v.1.1 criteria by investigators.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 24 months
  Progression free survival is defined as the time from the first day of serplulimab administration to progression disease or death，whichever occurs first, by the investigator according to Response Evaluation Criteria in Solid Tumors v.1.1 criteria or immune Response Evaluation Criteria in Solid Tumors v.1.1 criteria.
Overall Survival (OS) | Baseline up to approximately 36 months
  OS, defined as the time from initiation of study treatment to death from any cause. To assess clinical effectiveness of any serplulimab single used or combined therapy involved in this study by assessment of overall survival (OS) in patients with cervical Cancer. Time intervals for tumor assessment is every 6 or 12 week .
Duration of response (DOR) | Up to approximately 24 months
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time to the first disease progression | Up to approximately 24 months
  Ddefined as the interval between the date of the initial medication and the time of imaging progression.
1-year and 2-year Progression free survival Rate | Baseline up to approximately 24 months
  PFS is defined as the time from first administration to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PFS Rate was defined as the percentage of participants that are PFS event-free over 1-year and 2-year.
1-year and 2-year Overall Survival Rate | Baseline up to approximately 24 months
  OS, defined as the time from initiation of study treatment to death from any cause. OS Rate was defined as the percentage of participants that are OS event-free over 1-year and 2-year.
1-year and 2-year Disease Control Rate | Baseline up to approximately 24 months
  Percentage of all evaluable Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD) from first administration to 1-year and 2-year.

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD.PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No